CLINICAL TRIAL: NCT00475787
Title: Chiropractic Management of Chronic Lower Back Pain in Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CLIN-011-06F
Record Dates: First submitted 2007-05-17; First posted 2007-05-21 (Estimated); Results first posted 2014-12-30 (Estimated); Last update posted 2014-12-30 (Estimated); Status verified 2014-12

CONDITIONS: Chronic Low Back Pain
Keywords: Older Adults; Patient Education; Randomized Controlled Trial; Sham procedure; Spinal Manipulation; Veterans
MeSH Terms: interventions — Manipulation, Spinal

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Spinal Manipulative therapy (Experimental): Spinal manipulation involves high velocity low amplitude manipulation and flexion distraction and mobilization.
  Interventions: Procedure: Spinal Manipulation
- Detuned Ultrasound (Sham Comparator): Detuned Ultrasound involves utilizing an ultrasound machine that is set to "0 w/cm2" and US gel is applied to the spine for 11 minutes.
  Interventions: Procedure: Detuned Ultrasound

INTERVENTIONS:
Procedure: Spinal Manipulation — Spinal manipulation involves high velocity low amplitude manipulation and flexion distraction and mobilization.
  Arms: Spinal Manipulative therapy
Procedure: Detuned Ultrasound — US machine is turned on and set at "0 w/cm2"
  Other Names: Sham Procedure
  Arms: Detuned Ultrasound

SUMMARY:
The purpose of this study is to determine the effectiveness of Chiropractic management for treatment of chronic lower back pain in older adults.

DETAILED DESCRIPTION:
The identification of alternative safe and effective interventions for chronic lower back pain in the elderly is critical in view of its high prevalence, negative impact on quality of life and the treatment risks associated with chronic medication use. This is particularly germane to the veteran population, with a prevalence of lower back pain in excess of 40%. In 1998, published guidelines from the American Geriatric Society listed chiropractic management among the non-pharmacologic strategies for treating chronic pain symptoms in older adults. A recent study showed that a substantial number of older patients who received chiropractic care were less likely to be hospitalized, less likely to have used a nursing home, more likely to report a better health status, more likely to exercise vigorously and more likely to be mobile in the community. Patients undergoing chiropractic care have also reported greater satisfaction as compared to standard medical care. Despite the general clinical acceptance of chiropractic care and satisfaction with chiropractic services, evidence on the potential benefit and safety of chiropractic management of lower back pain in older adults is lacking. The purpose of this study is to evaluate the effectiveness of chiropractic management in older adults with chronic lower back pain, by comparing spinal manipulation to a sham intervention.

ELIGIBILITY:
Inclusion Criteria:

1. Pain greater than three months in duration
2. Localized pain to the lumbosacral and gluteal regions and no focal radicular symptoms
3. Pain elicited upon deep palpation of the lumbar erector spinae musculature 4) Pain that can be either exacerbated or relieved by varying body position

Exclusion Criteria:

1. Patients will be excluded if they have a history of fragility fracture of radiographic evidence of lumbar compression fracture
2. Patient will be excluded if they have undergone a course of previous chiropractic care
3. Severely demented patients, as indicated by their previous medical history and Mini Mental State scores of 22 or less, will not be selected.

   * The exclusion criteria are representative of the absolute contraindications for chiropractic management, specifically to mean high velocity, low amplitude spinal manipulation.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 136 (Actual)
Dates: Start 2008-04; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul Dougherty, DC, Principal Investigator — VA Medical Center, Canandaigua
Locations (2):
- United States (2):
  - VA Western New York Healthcare System at Buffalo, Buffalo, New York
  - VA Medical Center, Canandaigua, Canandaigua, New York

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm 1: Spinal manipulation involves high velocity low amplitude manipulation and flexion distraction and mobilization.
  Spinal Manipulation: Spinal manipulation involves high velocity low amplitude manipulation and flexion distraction and mobilization.
- Arm 2: Detuned Ultrasound
  Spinal Manipulation: Spinal manipulation involves high velocity low amplitude manipulation and flexion distraction and mobilization.
Period: Overall Study
Arm/Group | Arm 1 | Arm 2
Started | 69 | 67
Completed | 61 | 60
Not Completed | 8 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm 1 | Arm 2 | Total
Number analyzed (Participants) | 69 | 67 | 136
Age, Continuous [Mean (Standard Deviation); unit: years] | 77 (6.8) | 77 (6.81) | 77 (6.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2
  Male | 68 | 66 | 134

OUTCOME MEASURES:

1. Primary Outcome: Symptoms of Chronic Lower Back Pain as Measured With the Visual Analog Scale (VAS)
Description: 100 mm line with 0 being "no pain" and 100 mm being "the worst pain I can imagine".
Time Frame: Baseline, 5 weeks
Measure: Mean (95% Confidence Interval); unit: percentage of change from baseline to 5
Groups:
- Sham Group: Detuned Ultrasound
  Spinal Manipulation: Spinal manipulation involves high velocity low amplitude manipulation and flexion distraction and mobilization.
Arm/Group | Spinal Manipulative Therapy | Sham Group
Number analyzed (Participants) | 69 | 67
percentage of change from baseline to 5 | 26.32 [20.48 to 32.16] | 20.45 [14.18 to 26.71]

2. Secondary Outcome: Medical Outcome Study Short Form 36(SF-36) Bodily Pain
Description: For the Bodily pain subscale, the higher the number the less self-reported pain. The computed SF-36 pain subscale scores range from 2 to 12.
Time Frame: baseline and 5 Weeks
Measure: Mean (95% Confidence Interval); unit: percentage of change
Arm/Group | Arm 1 | Arm 2
Number analyzed (Participants) | 69 | 67
percentage of change | -1.01 [-1.42 to -.6] | -.53 [-.95 to -.11]

3. Secondary Outcome: Oswestry Disability Index (ODI)
Description: Validated measure of disability associated with lower back pain.
Time Frame: baseline and 5 weeks
Measure: Mean (95% Confidence Interval); unit: percentage of change
Arm/Group | Arm 1 | Arm 2
Number analyzed (Participants) | 69 | 67
percentage of change | 5.45 [2.82 to 8.07] | 3.42 [.08 to 6.04]

4. Secondary Outcome: Performance of the Timed up and go Test
Description: The Timed Up and Go Test assesses the amount of time it takes an individual to rise from a standard arm chair, walk a distance of 3 meters, and return to the initial position resting against the back of the chair, in this case the measurement was performed utilizing lasers to assess the time to the three meter mark and also the return to sitting in the chair.
Time Frame: baseline and 5 weeks
Measure: Mean (95% Confidence Interval); unit: percentage of change
Arm/Group | Arm 1 | Arm 2
Number analyzed (Participants) | 69 | 67
percentage of change | -1.17 [-2.11 to -.23] | -.65 [-1.39 to .09]

5. Secondary Outcome: Medical Outcome Study Short Form Physical Functioning Subscale
Description: For the Physical Functioning subscale, the higher the number the less self-reported limitations in physical function. The computed SF-36 physical function subscale scores range from 2 to 12.
Time Frame: baseline and 5 weeks
Measure: Mean (95% Confidence Interval); unit: percentage of change
Arm/Group | Spinal Manipulative Therapy | Sham Group
Number analyzed (Participants) | 69 | 67
percentage of change | -.06 [-.14 to .03] | -.05 [-015 to .04]

ADVERSE EVENTS:
Time Frame: Adverse event data were collected at each intervention/sham visit and at each of the data collection points (5 weeks, 12 weeks).
Description: Adverse event (AE) and serious adverse event (SAE) data were tracked for each group. An AE was defined as any undesirable medical event with new onset or significant exacerbation during the course of the study, regardless of whether or not it was considered to be related to study treatment.
Groups:
- Sham Intervention: Detuned Ultrasound
Arm/Group | Spinal Manipulative Therapy | Sham Intervention
Serious Adverse Events (participants affected / at risk) | 5/69 | 1/67
Other Adverse Events (participants affected / at risk) | 25/69 | 30/67
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Spinal Manipulative Therapy (N=69) | Sham Intervention (N=67)
Myelopathy (Nervous system disorders) | 1 (1) | 0 (0) — Patient was diagnosed with spondylotic myelopathy
Syncope (Cardiac disorders) | 2 (2) | 0 (0) — Cardiac related syncope, not related to study
myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1) — Unrelated MI
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — Patient fell on ice and injured lower back and neck
chest pain (Cardiac disorders) | 1 (1) | 0 (0) — Unrelated chest pain
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Spinal Manipulative Therapy (N=69) | Sham Intervention (N=67)
Back Pain (Musculoskeletal and connective tissue disorders) | 25/25 (50) | 30 (40)
Joint Pain (Musculoskeletal and connective tissue disorders) | 9 (11) | 13 (18)
leg pain (Musculoskeletal and connective tissue disorders) | 11 (18) | 4 (7)

LIMITATIONS AND CAVEATS:
1. Sham intervention was that it did involve some tactile stimulation
2. Only VA sites/predominantly male
3. Clinicians not blinded to invention delivered
4. All received educational booklet
5. Consideration of non-specific therapeutic effects

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes